CLINICAL TRIAL: NCT04906408
Title: The Effects of Post-Operative Interventions on Surgical Site Occurrences in Abdominal Wall Reconstructions: A Randomized Controlled Trial
Brief Title: The Effects of Post-Operative Interventions on Surgical Site Occurrences in AWR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Jeffrey Janis, Professor, Ohio State University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 2021H0061
Record Dates: First submitted 2021-05-18; First posted 2021-05-28 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Abdomen Hernia
Keywords: Infection; seroma; hematoma; skin necrosis; EC fistula; Mesh infection; Hernia recurrence; Bulge; Prevena; Prineo; Abdominal wall reconstruction; SSO; dressings
MeSH Terms: conditions — Hernia, Abdominal; Infections; Seroma; Hematoma; Necrosis

STUDY DESIGN:
Intervention Model Description: Partially blinded prospective, randomized-controlled trial
Who Masked: Investigator
Masking Description: Patient will not know what they received until randomization after consent process, surgeon will find out the day of surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Prevena (Experimental): Patients will then be randomized to group A (Prevena™) or group B (Prineo™) or group C (Standard wound dressing) using a random number generator made in Microsoft Excel. They will be made aware of which group they are in after the consent and randomization process, in order for proper post-operative teaching during the pre-operative clinic visit. The principal investigator, co-investigators and operating room staff will be aware of which post-operative intervention is being used on the day of surgery.
  Interventions: Device: Prevena
- Prineo (Experimental): Patients will then be randomized to group A (Prevena™) or group B (Prineo™) or group C (Standard wound dressing) using a random number generator made in Microsoft Excel. They will be made aware of which group they are in after the consent and randomization process, in order for proper post-operative teaching during the pre-operative clinic visit. The principal investigator, co-investigators and operating room staff will be aware of which post-operative intervention is being used on the day of surgery.
  Interventions: Device: Prineo
- Standard Dressing (Active Comparator): Patients will then be randomized to group A (Prevena™) or group B (Prineo™) or group C (Standard wound dressing) using a random number generator made in Microsoft Excel. They will be made aware of which group they are in after the consent and randomization process, in order for proper post-operative teaching during the pre-operative clinic visit. The principal investigator, co-investigators and operating room staff will be aware of which post-operative intervention is being used on the day of surgery.
  Interventions: Drug: Traditional

INTERVENTIONS:
Device: Prevena — Incisions will be dressed with closed incisional negative pressure wound therapy
  Arms: Prevena
Device: Prineo — Incisions will be dressed with Prineo
  Arms: Prineo
Drug: Traditional — Incisions will be dressed with bacitracin/xeroform
  Arms: Standard Dressing

SUMMARY:
Randomized controlled trial to compare SSO's in abdominal wall reconstruction patients using Prevena, Prineo, and traditional incisional dressings.

DETAILED DESCRIPTION:
Surgical site occurrences (SSOs) are a common complication of complex abdominal wall reconstruction (AWR), with rates ranging from 29-63.6%. Contributors to the high rates include: 1) comorbidities in this patient population such as; obesity, diabetes, smoking, and poor nutrition; 2) the need for complex surgical techniques including component separation, the use of mesh, skin resection, and the creation of adjacent skin flaps; 3) the possibility of contamination as a result of enterotomies or infected mesh from a previous procedure.

Any measures that can be taken to reduce the rates of surgical site occurrences are worthy of investigation, as they would help to decrease the morbidity and mortality of these procedures, while also potentially decreasing the overall cost associated with them. One measure of particular interest is what post-operative intervention, or wound dressing, is used. Many options exist. Those widely used include Prevena™, a vacuum assisted therapy that goes directly over the closed incision to assist with closure. This system works by placing a small piece of foam over the closed incision and then applying a vacuum over the foam. This allows the vacuum to apply uniformed pressure over the incision. It is thought that this vacuum creates negative pressure that helps to prevent contamination, hold the incision together, and remove fluid and infectious materials from the incision site. Another commonly used product is Prineo™, a self-adhering mesh that utilizes Dermabond™ glue technology that goes directly over the closed incision to assist with closure. The glue dries quickly over the incision and mesh, creating a barrier that is flexible but also resistant to contamination. While blocking potential contaminants such as water and bacteria from getting in, it allows water vapor to escape, while promoting a moist wound healing environment. There is also the traditional wound dressing which consists of Bacitracin antibiotics on a xeroform gauze, covered with a standard abdominal pad and tape.

Prevena™ has been widely studied in plastic surgery, specifically in AWR for large ventral hernias and for other complex abdominal reconstructions and is associated with reductions in SSOs from 22-51%. While there is strong evidence to support the use of Prevena in this patient population, there remains skepticism due to the lack of randomized, prospective studies to support its use. Prineo™ has not been studied as in depth, but multiple studies have shown it to be as efficacious as standard wound dressings in regard to wound healing, if not better.

There are currently no published reports comparing the rates of SSOs between these three therapies. This information is important to collect due to their potential abilities to reduce the rates of SSOs. Finding which decreases this rate the most can help guide decision making in our practice and potentially across the world.

When a patient with a ventral hernia or an abdominal wall tumor presents to the senior author for evaluation for abdominal wall reconstruction, a full history and physical examination will be performed. Patients who satisfy the study inclusion and exclusion criteria will be offered the opportunity to participate in the study. If they agree to participate, informed consent and HIPAA forms will be filled out and signed.

Patients will then be randomized to group A (Prevena™) or group B (Prineo™) or group C (Standard wound dressing) using a random number generator made in Microsoft Excel. They will not be told which group they are in, and only the principal investigator, co-investigators and operating room staff will be aware of which post-operative intervention is being used until after the surgery.

The patients will be asked to fill out 1 survey preoperatively: PROMIS Pain Intensity survey

They will then undergo surgery and will be followed within one week for wound dressing removal if needed, then at 6 weeks, 3 months, and 1 year and as needed. They will be evaluated for ventral hernia recurrence, bulge, or other SSOs throughout the follow-up period.

They will be asked to fill out the PROMIS Pain Intensity survey and POSAS 2.0 survey at 6 weeks, 3 months, and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Patients presenting for elective ventral hernia repair
* Patients deemed to be good surgical candidates, with no active life-threatening cardiac disease, pulmonary disease, renal disease, hematologic disease -Patients who will have a closed incision following the surgery

Exclusion Criteria:

* Known allergy to any material used in any wound treatment (Prevena- Acrylic adhesive or silver, Prineo- Dermabond glue, Standard- Bacitracin, Xeroform, surgical tape) -Active smokers (within the past 4 weeks) presenting for elective hernia repair
* Patients with active life-threatening cardiac disease, pulmonary disease, renal disease, hematologic disease presenting for elective ventral hernia repair
* Patients presenting for emergent ventral hernia repair (in the setting of bowel strangulation, necrosis, penetrating trauma) as it will be difficult to consent those patients for the study preoperatively
* Patients with severe systemic sepsis
* Patients with frank purulence in the wound -Patients with an open wound following surgery -Patients undergoing a panniculectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-09-17 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Infection | At 6 weeks postoperatively
Rate of Seroma | At 6 weeks postoperatively
Rate of Hematoma | At 6 weeks postoperatively
Rate of Dehiscence | At 6 weeks postoperatively
Rate of Skin necrosis | At 6 weeks postoperatively
Rate of Enterocutaneous fistula | At 6 weeks postoperatively
Rate of Mesh infection | At 6 weeks postoperatively
Rate of Hernia recurrence | At 6 weeks postoperatively
Rate of Bulge | At 6 weeks postoperatively

SECONDARY OUTCOMES:
Average Cost | At 6 weeks postoperatively
  In USD of postoperative wound care and complications
Average Cost | At 3 months postoperatively
  In USD of postoperative wound care and complications
Average Cost | At 1 year postoperatively
  In USD of postoperative wound care and complications
Average pain assessment score: PROMIS Pain Intensity survey | At 6 weeks postoperatively
  Minimum 3, Maximum 15, higher scores are worse pain/outcomes
Average pain assessment score: PROMIS Pain Intensity survey | At 3 months postoperatively
  Minimum 3, Maximum 15, higher scores are worse pain/outcomes
Average pain assessment score: PROMIS Pain Intensity survey | At 1 year postoperatively
  Minimum 3, Maximum 15, higher scores are worse pain/outcomes
Average scar assessment score: POSAS (Patient and Observer Scar) Assessment Scale) 2.0 survey | At 1 year postoperatively
  Provider score: Minimum 7, Maximum 70, higher scores are worse appearance/outcome.
  Patient score: Minimum 7, Maximum 70, higher scores are worse appearance/outcome.
Average scar assessment score: POSAS (Patient and Observer Scar) Assessment Scale) 2.0 survey | At 6 weeks postoperatively
  Provider score: Minimum 7, Maximum 70, higher scores are worse appearance/outcome.
  Patient score: Minimum 7, Maximum 70, higher scores are worse appearance/outcome.
Average scar assessment score: POSAS (Patient and Observer Scar) Assessment Scale) 2.0 survey | At 3 months postoperatively
  Provider score: Minimum 7, Maximum 70, higher scores are worse appearance/outcome.
  Patient score: Minimum 7, Maximum 70, higher scores are worse appearance/outcome.
Rate of infection | At 3 months postoperatively
Rate of infection | At 1 year postoperatively
Rate of Seroma | At 3 months postoperatively
Rate of Seroma | At 1 year postoperatively
Rate of Hematoma | At 1 year postoperatively
Rate of Hematoma | At 3 months postoperatively
Rate of Dehiscence | At 3 months postoperatively
Rate of Dehiscence | At 1 year postoperatively
Rate of Skin Necrosis | At 3 months postoperatively
Rate of Skin Necrosis | At 1 year postoperatively
Rate of Enterocutaneous fistula | At 3 months postoperatively
Rate of Enterocutaneous fistula | At 1 year postoperatively
Rate of Mesh infection | At 3 months postoperatively
Rate of Mesh infection | At 1 year postoperatively
Rate of Hernia Recurrence | At 3 months postoperatively
Rate of Hernia Recurrence | At 1 year postoperatively
Rate of Bulge | At 3 months postoperatively
Rate of Bulge | At 1 year postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey E Janis, MD, Principal Investigator — Ohio State University
Locations (1):
- Department of Plastic Surgery, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Not decided yet